CLINICAL TRIAL: NCT05386329
Title: Development and Preliminary Testing of a Non-regulated Digital Service That Supports Cognitive Behavioral Therapy for Depressive Symptoms Under Clinical Supervision
Brief Title: Therapist-Guided Smartphone-Delivered CBT for MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Koa Health B.V. (Industry)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Chief of Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P001958
Record Dates: First submitted 2022-04-19; First posted 2022-05-23 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: Digital Health; Cognitive Behavioral Therapy; Depression; Smartphone Apps; mHealth; Feasibility; Acceptability; Mobile App; Mental Health
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Interventional study without concurrent control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapist-guided smartphone-delivered CBT (Experimental): Participants will complete app-based cognitive-behavioral therapy (CBT) treatment for major depressive disorder (MDD) through their personal mobile smartphone. They will also be assigned a therapist, who will provide brief virtual treatment sessions (up to 25 minutes via a video platform) over the course of the same treatment period.
  Interventions: Behavioral: Mindset: Therapist-guided smartphone-delivered CBT

INTERVENTIONS:
Behavioral: Mindset: Therapist-guided smartphone-delivered CBT — All participants will receive the app-delivered CBT, including modules such as cognitive skills (e.g., cognitive restructuring, core belief work), behavioral skills (e.g., activity scheduling), and mindfulness. Therapists will also conduct brief weekly virtual appointments with participants.

SUMMARY:
We are testing a smartphone app that provides therapy for depression. Participants will also receive short weekly virtual appointments with a therapist. Researchers want to know if this new treatment is usable, whether participants are satisfied with it, and whether it can help lower symptoms.

DETAILED DESCRIPTION:
The purpose of this project is to conduct an open trial to test the feasibility, acceptability, and preliminary efficacy of a new therapist-guided smartphone-delivered cognitive behavioral therapy (CBT) for major depressive disorder (MDD). This treatment will include unlimited access to the mobile CBT for depression app over 8 weeks plus 8 virtual visits with a doctoral-level psychologist or psychology intern with their master's degree. The therapist will be assigned once eligibility is determined. All virtual sessions will be no longer than 16-25 min. The combined CBT app plus virtual treatment will be tested in 28 patients. Clinical assessments will occur at baseline, mid-treatment (week 4), end-of-treatment (week 8), and 3 month follow-up. The investigators hypothesize that this treatment will be feasible, acceptable to participants, and lead to reductions in depression symptoms and functional impairment as well as improvements in quality of life from baseline to end-of-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Living in Massachusetts
* Current primary diagnosis of depression
* at least moderately severe current symptoms of depression

Exclusion Criteria:

* Recent or anticipated changes in psychotropic medication use
* Past participation in a course of CBT for depression
* Current severe substance use disorder
* Lifetime bipolar disorder or psychosis
* Acute, active suicidal ideation
* Concurrent psychological treatment
* Does not own a supported mobile Smartphone with a data plan
* Lack of technology literacy that would interfere with ability to engage with smartphone treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bernstein EE, Daniel KE, Miyares PE, Hoeppner SS, Bentley KH, Snorrason I, Fisher LB, Greenberg JL, Weingarden H, Harrison O, Wilhelm S. Patterns of Skills Review in Smartphone Cognitive Behavioral Therapy for Depression: Observational Study of Intervention Content Use. JMIR Ment Health. 2025 Feb 24;12:e63497. doi: 10.2196/63497. PMID 39993308
- [Derived] Wilhelm S, Bernstein EE, Bentley KH, Snorrason I, Hoeppner SS, Klare D, Greenberg JL, Weingarden H, McCoy TH, Harrison O. Feasibility, Acceptability, and Preliminary Efficacy of a Smartphone App-Led Cognitive Behavioral Therapy for Depression Under Therapist Supervision: Open Trial. JMIR Ment Health. 2024 Apr 9;11:e53998. doi: 10.2196/53998. PMID 38592771

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapist-guided Smartphone-delivered CBT
Started | 28
End of Treatment | 26
Completed | 25
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Therapist-guided Smartphone-delivered CBT
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20
  Black | 1
  Asian/Pacific Islander | 3
  Other | 4
Region of Enrollment [Number; unit: participants]
  United States | 28
Sexual orientation [Count of Participants; unit: Participants]
  Straight or heterosexual | 20
  Bisexual | 5
  Lesbian, gay, or homosexual | 1
  Other | 2
Education [Count of Participants; unit: Participants]
  <= High school graduate | 4
  Technical school / some college | 5
  College graduate | 11
  Graduate or professional school | 8
Marital status [Count of Participants; unit: Participants]
  Single, never married | 19
  Married | 5
  Partnered | 2
  Separated / widowed | 2
Employment [Count of Participants; unit: Participants]
  Full-time (>= 35 h/wk) | 24
  Student | 2
  Unemployed | 1
  Retired | 1
Household income [Count of Participants; unit: Participants]
  $34,999 or less | 3
  $35,000 - 74,999 | 7
  $75,000 - 149,999 | 14
  $150,000 or more | 4
Geographic location [Count of Participants; unit: Participants]
  Urban | 12
  Suburban | 13
  Rural | 3
Duration of major depressive disorder (MDD), years [Mean (Standard Deviation); unit: years] | 15.5 (12.7)
Number of current comorbid MINI diagnoses [Count of Participants; unit: Participants]
  None | 15
  1 | 10
  2 | 0
  3 or more | 3

OUTCOME MEASURES:

1. Primary Outcome: Drop-Out Rates
Description: To determine feasibility, we will report rates of and reasons for participant dropout from the trial.
Time Frame: assessed at end-of-treatment (week 8)
Population: Data was analyzed in an intent to treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapist-guided Smartphone-delivered CBT
Number analyzed (Participants) | 28
Participants
  Lost contact | 2
  Completed treatment period | 26

2. Primary Outcome: Change in Patient Satisfaction (as Measured by the CSQ-8)
Description: The Client Satisfaction Questionnaire (CSQ) is an 8-item self-report questionnaire which assesses the satisfaction with clinical services received. Each item uses a 4-point Likert scale. Items are summed for a total score ranging from 8 to 32, with higher scores indicating greater satisfaction.
Time Frame: Measured at midpoint (week 4) and end-of-treatment (week 8)
Population: Data was analyzed in an intent to treat analysis with all people who completed questionnaires at week 4 (i.e., n=27/28). Data provided in the outcome measure data table are raw means from all available data, which includes missing data for one additional person who dropped out between week 4 and week 8.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist-guided Smartphone-delivered CBT
Number analyzed (Participants) | 27
score on a scale
  Week 4 | 26.3 (4.0)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 27.2 (3.3)
Statistical Analysis 1: Comparison: Therapist-guided Smartphone-delivered CBT; Null hypothesis: there is no significant difference in CSQ-8 total scores between midpoint (week 4) and end-of-treatment (week 8); Test type: Superiority — Comparison of mid-treatment to end-of-treatment; p = .0719, Mixed Models Analysis — The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with an unstructured covariance matrix; Mean Difference (Final Values) = 1.0308, 95% CI 2-sided [-0.09883 to 2.1605], Standard Error of Mean 0.5485 — The effect is presented as the therapist-guided smartphone-delivered CBT midpoint (week 4) CSQ-8 score compared to the end-point (week 8) CSQ-8 score

3. Primary Outcome: Change in Treatment Credibility (as Measured by the CEQ)
Description: The Credibility/Expectancy Questionnaire (CEQ) is a 6-item, self-report questionnaire. Items 1-3 assess clients' impressions of the treatment credibility; they are scored on Likert scales ranging from 1 to 9 (e.g., from 1='not at all' to 9='very much'). Items are summed for a total score that can range from 3 to 27, where higher scores mean greater treatment credibility.
Time Frame: Change in credibility from baseline (week 0) to midpoint (week 4)
Population: Data was analyzed in an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist-guided Smartphone-delivered CBT
Number analyzed (Participants) | 28
score on a scale
  Week 0 | 18.9 (3.1)
  Week 4: number analyzed (Participants) | 27
  Week 4 | 19.3 (3.8)
Statistical Analysis 1: Comparison: Therapist-guided Smartphone-delivered CBT; Null hypothesis: there is no significant difference in treatment credibility total scores between baseline (week 0) and midpoint (week 4); Test type: Superiority — Comparison of mid-treatment (week 4) to baseline; p = .6316, Mixed Models Analysis — The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with an unstructured covariance matrix; Mean Difference (Final Values) = 0.4296, 95% CI 2-sided [-1.3884 to 2.2475], Standard Error of Mean 0.8857 — The effect is presented as the therapist-guided smartphone-delivered CBT midpoint (week 4) CEQ credibility score compared to the baseline (week 0) CEQ credibility score

4. Primary Outcome: Change in Outcome Expectancy (as Measured by the CEQ)
Description: The Credibility/Expectancy Questionnaire (CEQ) is a 6-item, self-report questionnaire. Items 4-6 are used to assess clients' outcome expectancy. Item 5 is scored on a Likert scale ranging from 1 to 9 (where 1='not at all' to 9='very much'). Items 4 and 6 are scored on a scale from 0% to 100% (in 10-point increments); their scores are then converted linearly on a Likert scale from 1 to 9. Items are summed together for a total outcome expectancy score that can range from 3 to 27, where higher scores mean a higher outcome expectancy.
Time Frame: Measured at baseline (week 0) and midpoint (week 4)
Population: Data was analyzed in an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist-guided Smartphone-delivered CBT
Number analyzed (Participants) | 28
score on a scale
  Week 0 | 13.8 (3.3)
  Week 4: number analyzed (Participants) | 27
  Week 4 | 15.0 (5.4)
Statistical Analysis 1: Comparison: Therapist-guided Smartphone-delivered CBT; Null hypothesis: there is no significant difference in treatment expectancy total scores between baseline (week 0) and midpoint (week 4); Test type: Superiority — Comparison of mid-treatment (week 4) to baseline; p = .2225, Mixed Models Analysis — The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with an unstructured covariance matrix; Mean Difference (Final Values) = 1.1512, 95% CI 2-sided [-0.7422 to 3.0446], Standard Error of Mean 0.9213 — The effect is presented as the therapist-guided smartphone-delivered CBT midpoint (week 4) CEQ expectancy scores compared to the baseline (week 0) CEQ expectancy scores

5. Primary Outcome: App Rating (as Measured by the uMARS)
Description: The Mobile Application Rating Scale user version (uMARS) is a self-report form with 26 items that assess participant's evaluations of various app features. Dimensions of this measure include engagement (5 items), functionality (4 items), aesthetics (3 items), information quality (4 items); other items about app subjectivity quality (4 items) and perceived impact (6 items) are also available but do not contribute to the overall score (and are not reported here). Items are rated on differently worded 5-point Likert scales ranging from 1 (Inadequate) to 5 (Excellent). An overall app rating score can be calculated as the mean score of the first four subscales (engagement, functionality, aesthetics, and information quality; range of 1-5), where higher scores indicate higher overall perceived app quality.
Time Frame: Measured at endpoint (week 8)
Population: Data was analyzed from people who completed questionnaires at week 8 (i.e., n=26/28; "completers").
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist-guided Smartphone-delivered CBT
Number analyzed (Participants) | 26
units on a scale
  Engagement | 3.6 (0.6)
  Functionality | 4.5 (0.6)
  Aesthetics | 4.6 (0.5)
  Information quality | 4.6 (0.4)
  Overall app rating score | 4.3 (0.4)

6. Primary Outcome: Change in Treatment Utilization
Description: Treatment utilization was assessed with a single question: "On average, how much time (in minutes) do you spend using the app or practicing skills from the app in total, per week?" Answers were collected as number of minutes in integer format, where more time spent on and off the app was interpreted as greater treatment utilization.
Time Frame: Measured at midpoint (week 4) and end-of-treatment (week 8)
Population: Data was analyzed from people who completed questionnaires at week 4 (i.e., n=27/28), which was the first time this survey instrument was asked.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Therapist-guided Smartphone-delivered CBT
Number analyzed (Participants) | 27
minutes
  Week 4 | 50 [30 to 60]
  Week 8: number analyzed (Participants) | 26
  Week 8 | 60 [30 to 90]
Statistical Analysis 1: Comparison: Therapist-guided Smartphone-delivered CBT; Null hypothesis: There is no significant difference in treatment utilization between midpoint (week 4) and end of treatment (week 8); Test type: Superiority — Comparison of post-treatment (week 8) to mid-treatment (week 4); p = .7873, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was alpha=.05; Wilcoxon Z = 0.2712

7. Secondary Outcome: Change in MDD Symptom Severity (as Measured by the HAM-D)
Description: The Hamilton Depression Rating Scale (HAM-D) is the gold-standard clinician-administered assessment of depression symptom severity. It contains 21 items that are rated on a mixture of 3- and 5-point Likert scales. The first 17 items are summed for the total score, which can range from 0 to 52. Higher scores indicate greater depression severity.
Time Frame: Measured at baseline, week 4, week 8 (end of treatment), week 20 (follow-up)
Population: Data was analyzed in an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist-guided Smartphone-delivered CBT
Number analyzed (Participants) | 28
score on a scale
  Week 0 | 19.1 (5.0)
  Week 4: number analyzed (Participants) | 27
  Week 4 | 15.0 (6.1)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 10.8 (6.1)
  Week 20: number analyzed (Participants) | 25
  Week 20 | 9.8 (7.8)
Statistical Analysis 1: Comparison: Therapist-guided Smartphone-delivered CBT; Null hypothesis: there is no significant difference in HAM-D total scores between baseline (week 0) and end of treatment (week 8); Test type: Superiority — Pre-post comparison; p < .0001, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons because this was the pre-specified primary endpoint comparison. The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with an unstructured covariance matrix; Mean Difference (Final Values) = -7.8424, 95% CI 2-sided [-10.4944 to -5.1903], Standard Error of Mean 1.2858 — The effect is presented as the therapist-guided smartphone-delivered CBT end of treatment (week 8) HAM-D score compared to the baseline (week 0) HAM-D score

8. Secondary Outcome: Change in Functional Impairment (as Measured by the WSAS)
Description: The Work and Social Adjustment Scale (WSAS) is a self-report measure that assesses impairment in occupational, social, and family areas. The WSAS is a 5-item measure that uses 9-point Likert scales ranging from 0 (no impairment at all) to 8 (very severe impairment). The items are summed for a total score ranging from 0 to 40, where higher scores mean higher functional impairment.
Time Frame: Measured at baseline, week 4, week 8 (end of treatment), week 20 (follow-up)
Population: Data was analyzed in an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist-guided Smartphone-delivered CBT
Number analyzed (Participants) | 28
score on a scale
  Week 0 | 23.1 (7.8)
  Week 4: number analyzed (Participants) | 27
  Week 4 | 18.6 (7.9)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 13.0 (7.7)
  Week 20: number analyzed (Participants) | 25
  Week 20 | 12.3 (9.1)
Statistical Analysis 1: Comparison: Therapist-guided Smartphone-delivered CBT; Null hypothesis: there is no significant difference in WSAS total scores between baseline (week 0) and end of treatment (week 8); Test type: Superiority — Pre-post comparison; p < .0001, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons because this was the pre-specified secondary outcome that addresses complementary aspects of the patient experience. The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with an unstructured covariance matrix; Mean Difference (Final Values) = -9.9409, 95% CI 2-sided [-13.5043 to -6.3776], Standard Error of Mean 1.7329 — The effect is presented as the therapist-guided smartphone-delivered CBT end of treatment (week 8) WSAS scores compared to the baseline (week 0) WSAS scores

9. Secondary Outcome: Change in Quality of Life (as Measured by the Q-LES-Q-SF)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) is a 16-item, self-report questionnaire that assesses life satisfaction over the past week. Each question is rated on a 5-point Likert scale ranging from 1 (very poor) to 5 (very good). Questions 1-15 are then summed to a total score, and the total score is reported as a percentage maximum possible, such that the final percent score range is 0% to 100%, with higher scores indicating greater quality of life.
Time Frame: Measured at baseline, week 4, week 8 (end of treatment), week 20 (follow-up)
Population: Data was analyzed in an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist-guided Smartphone-delivered CBT
Number analyzed (Participants) | 28
score on a scale
  Week 0 | 40.9 (11.4)
  Week 4: number analyzed (Participants) | 27
  Week 4 | 52.4 (13.1)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 62.9 (13.5)
  Week 20: number analyzed (Participants) | 25
  Week 20 | 63.6 (14.3)
Statistical Analysis 1: Comparison: Therapist-guided Smartphone-delivered CBT; Null hypothesis: there is no significant difference in Q-LES-Q-SF total scores between baseline (week 0) and end of treatment (week 8); Test type: Superiority — Pre-post comparison; p < .0001, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons because this was a pre-specified secondary outcome assessing a complementary aspect of the patient experience. The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with an unstructured covariance matrix; Mean Difference (Final Values) = 21.5463, 95% CI 2-sided [14.5120 to 28.5806], Standard Error of Mean 3.4152 — The effect is presented as the therapist-guided smartphone-delivered CBT end of treatment (week 8) Q-LES-Q-SF percent scores compared to the baseline (week 0) Q-LES-Q-SF percent scores

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during study assessments at week 4, week 8, and the 3-month follow-up. At these assessments, participants were probed for adverse events that occurred since the last adverse event assessment.
Description: Participants were asked 4 questions about: (1) any major physical health problems or major physical injuries; (2) seeing a physical health or mental health provider for any reason; (3) any hospitalizations; or (4) any other major problems or concerns, all pertaining to the time since they were assessed last. Any "yes" resulted in a full event report. All serious adverse events are reported. Of non-serious events, only those affecting >5% in either treatment group are reported.
Arm/Group | Therapist-guided Smartphone-delivered CBT
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 18/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Therapist-guided Smartphone-delivered CBT (N=28)
Increased anxiety or depression (Psychiatric disorders) | 6
Suicidal ideation worsening (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 3
Bruising (Injury, poisoning and procedural complications) | 2
Other * (Infections and infestations) | 5 — * COVID-19, viral infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT05386329/Prot_SAP_000.pdf